CLINICAL TRIAL: NCT04860466
Title: A Phase 1, Multicenter, Open-label, Dose Finding Study of CC-96673 in Subjects With Relapsed or Refractory Non-Hodgkin's Lymphoma
Brief Title: A Dose Finding Study of CC-96673 in Participants With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-96673-NHL-001; 2020-004631-24 (EudraCT Number)
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-09

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Relapsed or Refractory; Non-Hodgkin's Lymphoma; CC-96673; Dose Finding
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of CC-96673 (Experimental): CC-96673 will be administered on a once weekly (Q1W) or once every 2 weeks (Q2W) schedule
  Interventions: Drug: CC-96673

INTERVENTIONS:
Drug: CC-96673 — IV Infusion

SUMMARY:
The purpose of this Phase 1 study is to evaluate the safety and tolerability of CC-96673 in adult participants with Relapsed or Refractory Non-Hodgkin's Lymphoma (R/R NHL).

The study will be conducted in 2 parts: Part A, monotherapy dose escalation and Part B, monotherapy dose expansion.

ELIGIBILITY:
Inclusion Criteria:

Participants must satisfy the following criteria to be enrolled in the study:

1. Participant (male or female) is ≥ 18 years of age at the time of signing the informed consent form (ICF).
2. Participant must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
3. Participant is willing and able to adhere to the study visit schedule and other protocol requirements.
4. Participant must have a history of NHL that has relapsed or progressed.
5. Participant has an ECOG PS of 0 or 1.
6. Participants must have acceptable laboratory values as specified in the protocol.

Exclusion Criteria:

1. Participant has cancer with symptomatic central nervous system (CNS) involvement
2. Participant is on chronic systemic immunosuppressive therapy or corticosteroids or subjects with clinically significant graft-versus-host disease (GVHD). Intranasal, inhaled, topical, or local corticosteroid injections, or steroids as premedication for hypersensitivity reactions are exceptions to this criterion.
3. Inadequate cardiac function or significant cardiovascular disease
4. Participant has received prior investigational therapy directed at CD47 or SIRPα.
5. Participant had major surgery ≤ 2 weeks prior to starting CC-96673.
6. Participant is a pregnant or lactating female or intends to become pregnant during participation of the study.
7. Participant has known active human immunodeficiency virus (HIV) infection.
8. Participant has active hepatitis B or C (HBV/HCV) infection.
9. Ongoing treatment with chronic, therapeutic dosing of anti-coagulants.
10. History of autoimmune hemolytic anemia or autoimmune thrombocytopenia.
11. History of concurrent second cancers requiring active, ongoing systemic treatment.
12. Participant has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
13. Participant has active, uncontrolled, or suspected infection. Other protocol defined inclusion/exclusion criteria could apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | From enrollment until at least 28 days after completion of study treatment
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a pre-existing condition) should be considered an AE.
Dose-limiting toxicity (DLT) | Up to approximately 18 months
  Number of participants with a DLT
Maximum tolerated dose (MTD) | Up to approximately 18 months
  Is defined as the dose level that can be given such that the estimated DLT probability is closest to approximately 30%.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years after study treatment
  Is defined as the percent of participants whose best response is CR or PR
Time to response (TTR) | Up to 2 years after study treatment
  Is defined as the time from the first dose of CC-96673 to tumor response
Duration of response (DOR) | Up to 2 years after study treatment
  Is defined as the time from tumor response to progression/death
Progression free survival (PFS) | Up to 2 years after study treatment
  Is defined as the time from the first dose of CC-96673 to the first occurrence of disease progression or death from any cause
Pharmacokinetics - Cmax | Up to 24 Months
  Maximum observed serum concentration of drug
Pharmacokinetics - AUC | Up to 24 Months
  Area under the serum concentration-time curve
Pharmacokinetics - tmax | Up to 24 Months
  Time of maximum observed serum concentration
Incidence of laboratory-reported positive responses of anti-CC-96673 antibodies | Up to 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (13):
- United States (4):
  - Local Institution - 104, Minneapolis, Minnesota
  - Local Institution - 103, Omaha, Nebraska
  - Local Institution - 101, Houston, Texas
  - Local Institution - 102, Seattle, Washington
- Canada (2):
  - Local Institution - 201, Toronto, Ontario
  - Local Institution - 202, Montreal, Quebec
- France (4):
  - Local Institution - UNK-5, Angers
  - Local Institution - 303, Lille
  - Local Institution - 302, Montpellier
  - Hopital Lyon Sud, Pierre-Bénite
- Spain (3):
  - Local Institution - 401, Madrid
  - Local Institution - 403, Málaga
  - Local Institution - 402, Salamanca

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com